CLINICAL TRIAL: NCT00724022
Title: Triple Arm, Prospectively Randomized Multi Centre Study Phase IV to Evaluate Calcineurin Inhibitor Reduced, Steroid Free Immunosuppression After Renal Transplantation in Non-risk Patients
Brief Title: Phase IV Study to Evaluate Calcineurin Inhibitor Reduced, Steroid Free Immunosuppression After Renal Transplantation
Acronym: Harmony
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Collaborators: Roche Pharma AG (Industry); Astellas Pharma GmbH (Industry); Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Prof. Dr.med. Oliver Thomusch, Professor, University Hospital Freiburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IT1850071; EudraCT No. 2007-006516-31; DRKS00000452 (Registry Identifier: German Clinical Trials Register)
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Disorder Related to Renal Transplantation
Keywords: Kidney transplant status; Steroid free; Reduced; Calcineurin; Inhibitor; Immunosuppression
MeSH Terms: interventions — Basiliximab; Tacrolimus; Mycophenolic Acid; Prednisone; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Other): Standard: Advagraf, CellCept, Decortin H + 2x Simulect Day 0 + 4
  Interventions: Drug: Basiliximab, Tacrolimus, MMF, Prednisolon
- B (Experimental): Steroidfree: Advagraf, Cellcept, Decortin H until Day 8, 2x Simulect Day 0 + 4
  Interventions: Drug: Basiliximab, Tacrolimus, MMF
- C (Experimental): Steroidfree: Advagraf, Cellcept, Decortin H until Day 8, 3 x Thymoglobulin
  Interventions: Drug: Tacrolimus, MMF, rATG

INTERVENTIONS:
Drug: Basiliximab, Tacrolimus, MMF, Prednisolon — Control group. Therapy with Prednisolon.
  Other Names: Simulect; Advagraf; CellCept; Decortin
  Arms: A
Drug: Basiliximab, Tacrolimus, MMF — No Prednisolon after 7 days
  Other Names: Simulect; Advagraf; CellCept
  Arms: B
Drug: Tacrolimus, MMF, rATG — Induction therapy: rATG instead of Basiliximab. No Prednisolon.
  Other Names: Advagraf; CellCept; Thymoglobulin
  Arms: C

SUMMARY:
Current practice of immune suppressive standard therapy after renal transplantation in non-risk patients is a triple therapy consisting of steroids, a calcineurin inhibitor and MMF. The aim of this clinical trial is to combine a reduction of CNI using tacrolimus and a concept of not using steroids in order to establish an immunosuppressive regimen in immunologically non-risk patients that is efficient and causes as few side effects as possible.

DETAILED DESCRIPTION:
In this triple arm, prospectively randomized multi centre phase IV study 200 patients per study arm will be investigated for 12 months.

Based on the results of the Symphony study the low dose tacrolimus study arm will be modified to further improve efficacy (prevention of BPAR, best possible renal function) and safety (adverse event profile regarding infections, cardiovascular risk factors, malignant tumours) of immunosuppression. For this, CNI will be reduced and in addition the rate of steroid free patients after 1 week will be maximized to achieve a long lasting improved post surgical cardiovascular risk profile (in particular concerning de novo induction of diabetes mellitus and other adverse events caused by steroids). Safety should be increased without loss of efficacy of immunosuppression (measured in rejection rate and allograft loss rate) as compared to an immune suppressive therapy comprising steroids. Therefore, following the successful study arm of the Symphony study, immunosuppression in the first of the three study arms comprises a steroid in combination with Advagraf and CellCept in addition to a two dose induction therapy with Simulect (group A). The regimen of the second study arm is similar but discontinues steroids on day seven after transplantation (group B). Therapy of group three is similar to group B but Simulect is replaced by T-cell depleting polyclonal antibodies (Thymoglobulin) (group C).

ELIGIBILITY:
Inclusion Criteria:

* Post mortal kidney donation or living donation
* Primary and secondary renal transplantation, unless the graft was lost due to severe rejection within the first year
* PRA level ≤ 20%.
* Recipient ≥ 18 to 75 years of age
* AB0-compatible
* Negative crosshatch
* Patients with a signed informed consent form
* Women of child-bearing age must agree to an efficient contraception

Exclusion Criteria:

* Third or multiple transplantation
* Transplantation per a "non-heart beating" donor
* HLA-identical living donation
* Incompatibility to study medication (allergy, intolerance, hypersensitivity)
* Patients with existing malignant underlying disease or tumour anamnesis < 5 years. Exception: basaloma or squamous cell carcinoma of the skin after successful therapy
* Female patients who do not use a safe method of contraception
* Patients with clinically significant, uncontrolled infectious diseases (incl. HIV) and/or severe diarrhoea, emesis, active malabsorption of the upper gastrointestinal tract or active peptic ulcer
* Patients currently, resp. within the last 30 days, participating in other studies
* Primary focal-sclerosing glomerulonephritis and membranoproliferative glomerulonephritis as an underlying disease
* Autoimmune disease as underlying disease (collagen diseases, colitis, HUS, SLE) which might require chronic cortisone therapy
* Additional disease requiring temporary or chronic cortisone therapy (including inhalation medicine)
* Chronic hepatitis B and hepatitis C infection
* Thrombopenia < 70.000/mm3 or leukopenia < 2.500/mm3 or neutropenia < 1500/ mm3.
* Patients with hepatocirrhosis Child B or C or another severe disease of the liver
* Patients with symptoms of a significant somatic or psychiatric / mental illness. Patients who are not able to realize nature, relevance and consequences of the clinical trial and who are not able to comply, to cooperate and communicate adequately and to follow the instructions of the study or even to give their informed consent (according to § 40 article 4 and § 41 article 2 and 3 AMG).
* Patients who possibly depend on the sponsor or the trial physician
* Patients with signs of drug abuse or alcohol abuse
* Patients taking additional medicines with known interactions with the immune suppressive substances (MMF and tacrolimus) that preclude an adequate control of the immunosuppression
* Cold ischemia time of donor kidney > 30 hours
* Pregnant or nursing patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2008-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Efficacy of immunosuppression measured in rejection rate confirmed by biopsy according to BANFF 97, modified 2005. | one year after transplantation

SECONDARY OUTCOMES:
Rate of patients with steroid-free immunosuppression
  Rate of patients with steroid-free immunosuppression
patient and graft survival rate
  patient and graft survival rate
graft function (calculated by the Cock- croft-Gault and MDRD-IV formula respectively calculated creatinine clearance by the Nankivell formula respectively cystatin C measurement)
  graft function (calculated by the Cock- croft-Gault and MDRD-IV formula respectively calculated creatinine clearance by the Nankivell formula respectively cystatin C measurement)
Number of steroid-resistant rejections
  Number of steroid-resistant rejections
blood pressure level and also amount and types of blood pressure medications
  blood pressure level and also amount and types of blood pressure medications
Lipid levels and also amount and types of lipid-lowering medications
  Lipid levels and also amount and types of lipid-lowering medications
body weight, relative weight gain [kg], BMI
  body weight, relative weight gain [kg], BMI
infection rate, infection type and infection severity
  infection rate, infection type and infection severity
anemia requiring erythropoietin treatment
  anemia requiring erythropoietin treatment
PTLD incidence
  PTLD incidence
tumor incidence
  tumor incidence
incidence of diabetes mellitus nd incidence of abnormal fasting blood sugar levels respectively incidence of impaired glucose tolerance, incidence of de novo insulin-requiring or oral-antidiabetic-requiring treatment over ≥30 days | 30 days
  incidence of diabetes mellitus (ADA criteria, venous blood glucose concentration on an empty stomach ≥7.0 mmol/l, pathologic OGTT) and incidence of abnormal fasting blood sugar levels respectively incidence of impaired glucose tolerance, incidence of de novo insulin-requiring or oral-antidiabetic-requiring treatment over ≥30 days
incidence of cataracts
  incidence of cataracts
incidence of avascular necrosis
  incidence of avascular necrosis
incidence of osteoporosis
  incidence of osteoporosis (assessment of fracture rate, osteodensitometry)
Wound healing disorders
  Wound healing disorders
incidence of chronic allograft nephropathy (CAN) (12-month histology)
  incidence of chronic allograft nephropathy (CAN) (12-month histology)
incidence of CMV disease (qPCR >1000 copies/μL)
  incidence of CMV disease (qPCR >1000 copies/μL)
incidence of BKV disease (qPCR >1000 copies/μL)
  incidence of BKV disease (qPCR >1000 copies/μL)
incidence of EBV disease (qPCR >1000 copies/μL)
  incidence of EBV disease (qPCR >1000 copies/μL)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Hopt, Prof.Dr.Dr., Study Director — University Hospital Freiburg; Oliver Thomusch, Prof. Dr., Principal Investigator — University Hospital Freiburg; Christian Hugo, Prof. Dr., Principal Investigator — Universitaetsklinikum Erlangen
Locations (25):
- Germany (25):
  - Universitaetsklinikum Berlin, Berlin
  - Universitaetsklinikum Bonn, Bonn
  - Klinikum Bremen-Mitte, Bremen
  - Universitaetsklinikum Koeln, Cologne
  - Kliniken der Stadt Köln gGmbH - Krankenhaus Köln-Merheim, Cologne
  - Carl Gustav Carus Universitätsklinikum, Dresden
  - Universitaetsklinikum Erlangen, Erlangen
  - Universitaetsklinikum Essen, Essen
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Nephrologisches Zentrum Niedersachsen, Hannoversch Münden
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Jena, Jena
  - Transplantationszentrum Kaiserslautern, Kaiserslautern
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum Schleswig-Holstein Campus Lübeck, Lübeck
  - Universitätsklinikum Mainz, Mainz
  - Universitaetsklinikum Mannheim, Mannheim
  - Universitätsklinikum München LMU, München
  - Klinikum rechts der Isar der TU München, München
  - Universitaetsklinikum der WWU Münster, Münster
  - Universitätsklinikum Regensburg, Regensburg
  - Universitätsklinikum Rostock, Rostock
  - Universitätsklinikum Tübingen, Tübingen
  - Universitaetsklinikum Würzburg, Würzburg

REFERENCES:
- [Derived] Wajih Z, Karpe KM, Walters GD. Interventions for BK virus infection in kidney transplant recipients. Cochrane Database Syst Rev. 2024 Oct 9;10(10):CD013344. doi: 10.1002/14651858.CD013344.pub2. PMID 39382091
- [Derived] Stumpf J, Thomusch O, Opgenoorth M, Wiesener M, Pascher A, Woitas RP, Suwelack B, Rentsch M, Witzke O, Rath T, Banas B, Benck U, Sommerer C, Kurschat C, Lopau K, Weinmann-Menke J, Jaenigen B, Trips E, Hugo C. Excellent efficacy and beneficial safety during observational 5-year follow-up of rapid steroid withdrawal after renal transplantation (Harmony FU study). Nephrol Dial Transplant. 2023 Dec 20;39(1):141-150. doi: 10.1093/ndt/gfad130. PMID 37391381
- [Derived] Wittenbrink N, Herrmann S, Blazquez-Navarro A, Bauer C, Lindberg E, Wolk K, Sabat R, Reinke P, Sawitzki B, Thomusch O, Hugo C, Babel N, Seitz H, Or-Guil M. A novel approach reveals that HLA class 1 single antigen bead-signatures provide a means of high-accuracy pre-transplant risk assessment of acute cellular rejection in renal transplantation. BMC Immunol. 2019 Apr 27;20(1):11. doi: 10.1186/s12865-019-0291-2. PMID 31029086
- [Derived] Thomusch O, Wiesener M, Opgenoorth M, Pascher A, Woitas RP, Witzke O, Jaenigen B, Rentsch M, Wolters H, Rath T, Cingoz T, Benck U, Banas B, Hugo C. Rabbit-ATG or basiliximab induction for rapid steroid withdrawal after renal transplantation (Harmony): an open-label, multicentre, randomised controlled trial. Lancet. 2016 Dec 17;388(10063):3006-3016. doi: 10.1016/S0140-6736(16)32187-0. Epub 2016 Nov 19. PMID 27871759